CLINICAL TRIAL: NCT04635748
Title: Feasibility of Collateral Information Review and Its Impact on Clinical Decision-Making
Status: Completed | Type: Observational
Sponsor: Mclean Hospital (Other)
Collaborators: Once Upon a Time Foundation (Other)
Responsible Party: Principal Investigator, Ipsit Vihang Vahia, Medical Director, Geriatric Psychiatry Outpatient Services, Mclean Hospital
Other Study IDs: 2019P003450
Record Dates: First submitted 2020-11-13; First posted 2020-11-19 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Depressive Disorder; Anxiety Disorders
MeSH Terms: conditions — Depressive Disorder; Anxiety Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This project will investigate how review of collateral information sources (CIS) may impact clinical decision-making across the lifespan.

DETAILED DESCRIPTION:
This study aims to explore how reviewing collateral information sources (CIS) may affect clinical decision-making for clinicians treating participants with varied mood disorders. Investigators will assess the types of collateral information used in the clinical setting and treatment decisions made after a clinical session. We will gather this information from interested clinicians who will provide this information after each patient visit over the course of one week.

ELIGIBILITY:
Inclusion Criteria:

1. Credentialed to provide psychopharmacology or psychotherapy at McLean and Licensed by the State of Massachusetts
2. Practice pharmacotherapy and either adjunctive or stand-alone evidence-based psychotherapy (e.g., CBT, DBT, supportive psychotherapy, etc.)
3. Fluent in English

Exclusion Criteria:

* Clinicians who do not meet the inclusion criteria detailed above

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: - Clinicians from McLean Hospital Outpatient Programs (geriatric, child and adult) and the McLean Behavioral Health Partial Program, which predominantly treat patients with mood disorders.
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2019-12-03 (Actual); Primary Completion 2020-03-14 (Actual); Study Completion 2020-03-14 (Actual)

PRIMARY OUTCOMES:
McLean Treatment Tracking Survey | Over the course of 1 week
  Clinicians will find the McLean Treatment Tracking Survey easy to use in their clinical care and we will measure rate of use and completion.

SECONDARY OUTCOMES:
Clinical Outcome - Increased treatment decisions made | Over the course of 1 week
  Investigators will explore whether reviewing more collateral information sources leads to more clinical actions taken for treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Ipsit V Vahia, MD, Principal Investigator — Mclean Hospital; Kerry J Ressler, MD; PhD, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States